CLINICAL TRIAL: NCT05398887
Title: Utilization and Effectiveness of Ultra-low-dose Chest Computed Tomography Using Innovative CT Denoising Solution Based on Deep Learning Technology
Brief Title: Effectiveness of Ultra-low-dose Chest CT With AI Based Denoising Solution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Intermed Hospital (Other)
Responsible Party: Principal Investigator, Bayarbaatar Bold, Principal Investigator, Bayarbaatar Bold, Diagnostic Radiologist, M.D, Intermed Hospital, Intermed Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: IMC20220515-01
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Lung Diseases
Keywords: Computed tomography; Artificial Intelligence; Denoising technique; Ultra-low-dose Computed tomography
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose Chest CT scan (Active Comparator): Underwent low dose chest CT with 30% lower radiation dose
  Interventions:
  Radiation: Low radiation dose CT Other: Image quality analysis
  Interventions: Radiation: Low radiation dose CT
- Ultra low dose CT scan with Artificial Intelligence (Experimental): Interventions:
  Radiation: Low radiation dose CT Image quality Other: Deep-learning based contrast boosting algorithms
  Interventions: Radiation: Underwent ultra dose chest CT; Other: Artificial Intelligence based model

INTERVENTIONS:
Radiation: Low radiation dose CT — Underwent low dose chest CT with 30% lower radiation dose
  Arms: Low dose Chest CT scan
Radiation: Underwent ultra dose chest CT — Underwent ultra dose chest CT with 90% lower radiation dose
  Arms: Ultra low dose CT scan with Artificial Intelligence
Other: Artificial Intelligence based model — Deep-learning based contrast boosting algorithms
  Arms: Ultra low dose CT scan with Artificial Intelligence

SUMMARY:
The main objective of the study is to evaluate the detection rate of pulmonary conditions, percentage of ionizing radiation dose reduction, and state of image quality of ULDCT coupling with innovative vendor-neutral CT denoising solution based on deep learning technology.

DETAILED DESCRIPTION:
Considering lung cancer-related public health challenges, a reliable lung cancer screening method for high-risk cohorts in Mongolia is needed. Thus, our study aims to assess the detection rate of pulmonary conditions, percentage of ionizing radiation dose reduction, and state of image quality of ULDCT coupling with artificial intelligence based CT denoising technique among various patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18-year-old
* Patients undergoing CT Chest for all purpose

Exclusion Criteria:

* Age less than 18 years
* Any suspicion of pregnancy
* History of thoracic surgery or placement of the metallic device in the thorax
* An inability to hold respiration during CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of pulmonary conditions | Within 2 weeks after data collection
  Pulmonary condition detection rate on low dose chest CT and ultra dose chest CT with artificial intelligence-based CT denoising solution by blinded reviewers
Contrast media dose | Within 2 weeks after data collection
  Administered contrast media dose in each patient

SECONDARY OUTCOMES:
Image contrast | Within 2 weeks after data collection
  Signal to Noise, Noise and Edge-rise-distance on a five-point scale (1-5) with a higher score indicates better conspicuity.

CONTACTS AND LOCATIONS:
Overall Officials: Khulan Khurelsukh, M.D, MSc, Study Chair — Intermed Hospital; Delgerekh Sainjargal, M.D, MSc, Principal Investigator — Intermed Hospital; Bayarbaatar Bold, M.D, Principal Investigator — Intermed Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] International Agency for Research on Cancer. Global Cancer Observatory: cancer today. World Health Organization. https://gco.iarc.fr/today (accessed Feb 14, 2022).
- [Background] Health Development Center, WHO. Health Indicators 2019. Mongolian Health Development Center. http://hdc.gov.mn/media/uploads/202108/Eruul_mendiin_uzuulelt_2020.pdf (accessed Feb 14, 2022).
- [Background] WHO global report. WHO global report on mortality attributable to tobacco. 2012
- [Background] Zheng W, McLerran DF, Rolland BA, Fu Z, Boffetta P, He J, Gupta PC, Ramadas K, Tsugane S, Irie F, Tamakoshi A, Gao YT, Koh WP, Shu XO, Ozasa K, Nishino Y, Tsuji I, Tanaka H, Chen CJ, Yuan JM, Ahn YO, Yoo KY, Ahsan H, Pan WH, Qiao YL, Gu D, Pednekar MS, Sauvaget C, Sawada N, Sairenchi T, Yang G, Wang R, Xiang YB, Ohishi W, Kakizaki M, Watanabe T, Oze I, You SL, Sugawara Y, Butler LM, Kim DH, Park SK, Parvez F, Chuang SY, Fan JH, Shen CY, Chen Y, Grant EJ, Lee JE, Sinha R, Matsuo K, Thornquist M, Inoue M, Feng Z, Kang D, Potter JD. Burden of total and cause-specific mortality related to tobacco smoking among adults aged >/= 45 years in Asia: a pooled analysis of 21 cohorts. PLoS Med. 2014 Apr 22;11(4):e1001631. doi: 10.1371/journal.pmed.1001631. eCollection 2014 Apr. PMID 24756146
- [Background] Fourth national STEPS Survey on the Prevalence of Noncommunicable Disease and Injury Risk Factors-2019. World Health Organization.
- [Background] Smith-Bindman R, Lipson J, Marcus R, Kim KP, Mahesh M, Gould R, Berrington de Gonzalez A, Miglioretti DL. Radiation dose associated with common computed tomography examinations and the associated lifetime attributable risk of cancer. Arch Intern Med. 2009 Dec 14;169(22):2078-86. doi: 10.1001/archinternmed.2009.427. PMID 20008690
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] Boyd MA. U.S. radiation protection: role of national and international recommendations and opportunities for collaboration (harmony, not dissonance). Health Phys. 2015 Feb;108(2):278-82. doi: 10.1097/HP.0000000000000236. PMID 25551510
- [Background] Katsura M, Matsuda I, Akahane M, Yasaka K, Hanaoka S, Akai H, Sato J, Kunimatsu A, Ohtomo K. Model-based iterative reconstruction technique for ultralow-dose chest CT: comparison of pulmonary nodule detectability with the adaptive statistical iterative reconstruction technique. Invest Radiol. 2013 Apr;48(4):206-12. doi: 10.1097/RLI.0b013e31827efc3a. PMID 23344517
- [Background] Kim Y, Kim YK, Lee BE, Lee SJ, Ryu YJ, Lee JH, Chang JH. Ultra-Low-Dose CT of the Thorax Using Iterative Reconstruction: Evaluation of Image Quality and Radiation Dose Reduction. AJR Am J Roentgenol. 2015 Jun;204(6):1197-202. doi: 10.2214/AJR.14.13629. PMID 26001228
- [Background] Lee SW, Kim Y, Shim SS, Lee JK, Lee SJ, Ryu YJ, Chang JH. Image quality assessment of ultra low-dose chest CT using sinogram-affirmed iterative reconstruction. Eur Radiol. 2014 Apr;24(4):817-26. doi: 10.1007/s00330-013-3090-9. Epub 2014 Jan 18. PMID 24442444
- [Background] Nagatani Y, Takahashi M, Murata K, Ikeda M, Yamashiro T, Miyara T, Koyama H, Koyama M, Sato Y, Moriya H, Noma S, Tomiyama N, Ohno Y, Murayama S; investigators of ACTIve study group. Lung nodule detection performance in five observers on computed tomography (CT) with adaptive iterative dose reduction using three-dimensional processing (AIDR 3D) in a Japanese multicenter study: Comparison between ultra-low-dose CT and low-dose CT by receiver-operating characteristic analysis. Eur J Radiol. 2015 Jul;84(7):1401-12. doi: 10.1016/j.ejrad.2015.03.012. Epub 2015 Apr 2. PMID 25892051
- [Background] Wang R, Sui X, Schoepf UJ, Song W, Xue H, Jin Z, Schmidt B, Flohr TG, Canstein C, Spearman JV, Chen J, Meinel FG. Ultralow-radiation-dose chest CT: accuracy for lung densitometry and emphysema detection. AJR Am J Roentgenol. 2015 Apr;204(4):743-9. doi: 10.2214/AJR.14.13101. PMID 25794063
- [Background] Yanagawa M, Gyobu T, Leung AN, Kawai M, Kawata Y, Sumikawa H, Honda O, Tomiyama N. Ultra-low-dose CT of the lung: effect of iterative reconstruction techniques on image quality. Acad Radiol. 2014 Jun;21(6):695-703. doi: 10.1016/j.acra.2014.01.023. Epub 2014 Apr 6. PMID 24713541
- [Background] Tsushima E. Intraclass correlation coefficient as a reliability index [Japanese]. http://www.hs.hirosaki-u.ac.jp/~pteiki/research/stat/icc.pdf. Accessed 9 Feb 2017.
- [Background] Svahn TM, Sjoberg T, Ast JC. Dose estimation of ultra-low-dose chest CT to different sized adult patients. Eur Radiol. 2019 Aug;29(8):4315-4323. doi: 10.1007/s00330-018-5849-5. Epub 2018 Dec 17. PMID 30560356
- [Background] Afadzi M, Fossa K, Andersen HK, Aalokken TM, Martinsen ACT. Image Quality Measured From Ultra-Low Dose Chest Computed Tomography Examination Protocols Using 6 Different Iterative Reconstructions From 4 Vendors, a Phantom Study. J Comput Assist Tomogr. 2020 Jan/Feb;44(1):95-101. doi: 10.1097/RCT.0000000000000947. PMID 31939889
- [Background] Zhang M, Qi W, Sun Y, Jiang Y, Liu X, Hong N. Screening for lung cancer using sub-millisievert chest CT with iterative reconstruction algorithm: image quality and nodule detectability. Br J Radiol. 2018 Oct;91(1090):20170658. doi: 10.1259/bjr.20170658. Epub 2017 Dec 5. PMID 29120665